CLINICAL TRIAL: NCT02671721
Title: Intraoperative Protective Ventilation and Postoperative Pulmonary Complications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Mayo Clinic (Other); University of Colorado, Denver (Other)
Responsible Party: Principal Investigator, Marcos Vidal Melo, MD, PhD, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2015P001613
Record Dates: First submitted 2016-01-30; First posted 2016-02-02 (Estimated); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Complication of Ventilation Therapy; Postoperative Respiratory Complications

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional Strategy (No Intervention): Patients will receive usual and prudent PEEP and tidal volume settings.
- Maximal Compliance Strategy (Experimental): PEEP will be set at the maximum static respiratory system compliance during a descending PEEP titration curve.
  Interventions: Other: Maximal Compliance
- Transpulmonary Pressure Strategy (Experimental): Personal PEEP titration using transpulmonary pressures obtained from a naso/orogastric tube containing an esophageal balloon port
  Interventions: Other: Transpulmonary Pressure

INTERVENTIONS:
Other: Maximal Compliance — PEEP will be set at the maximum static respiratory system compliance during a descending PEEP titration curve.
  Arms: Maximal Compliance Strategy
Other: Transpulmonary Pressure — We will use transpulmonary pressure values obtained using an naso/orogastric tube during the operative procedure to titrate PEEP intraoperatively.
  Arms: Transpulmonary Pressure Strategy

SUMMARY:
The purpose of this pilot study is to identify the optimal way to ventilate patients during abdominal surgery in order to reduce the amount of post-operative pulmonary complications in patients at moderate and high-risk for them.

DETAILED DESCRIPTION:
The investigators plan to prospectively compare two methods to individualize Positive End Expiratory Pressure (PEEP) settings in the operating room during abdominal surgery: (1) Maximization of respiratory compliance during a decremental PEEP titration, and (2) Prevention of negative end-expiratory transpulmonary pressures.

The investigators will exploit the usual intraoperative requirement for a naso/orogastric tube to assess transpulmonary pressures,and respiratory mechanics measurements from anesthesia machines to titrate PEEP.

The investigators will measure biomarkers of lung injury and lung function to compare those methods between themselves and to the control group. In the process, the investigators will assess the ease and reliability of anesthesia teams in implementing the methods. These data will allow us to determine the PEEP strategy best suited for the full-scale trial, and to estimate the degree of separation the experimental lung protective approach will have from the protocolized usual care control settings.

ELIGIBILITY:
Inclusion Criteria:

* Adults ( 18 years) scheduled for elective surgery expected to last 2 h,
* elective intraperitoneal abdominal or pelvic surgery including: gastric; biliary; pancreatic; hepatic; major bowel, ovarian, renal tract, bladder, and prostatic; radical hysterectomy; and pelvic exenteration;
* at least intermediate risk of PPCs defined by a risk score 26

Exclusion Criteria:

* Inability or refusal to provide consent
* Refusal of clinicians caring for patient to follow the protocol
* Participation in interventional investigation within 30 days of the time of the study
* Pregnancy
* Emergency surgery
* Severe obesity (above Class I, BMI 35)
* Significant lung disease: any diagnosed or treated respiratory condition that (a) requires home oxygen therapy or non-invasive ventilation, (b) severely limits exercise tolerance to <4 METs (e.g. patients unable to do light housework, walk flat at 4 miles/h or climb one flight of stairs), or (c) required previous lung surgery80
* Significant heart disease: cardiac conditions that limit exercise tolerance to <4 METs
* Renal failure: peritoneal or hemodialysis requirement or preoperative creatinine 2 mg/dL;
* Neuromuscular disease that impairs ability to ventilate without assistance
* Severe chronic liver disease (Child-Pugh Score of 10 -15)
* Sepsis
* Malignancy or other irreversible condition for which 6-month mortality is estimated 50%
* Bone marrow transplant.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Intraoperative driving pressure | During abdominal surgery
  We will assess intraoperative driving pressure to evaluate respiratory mechanics during surgery.
Intraoperative transpulmonary pressure | During abdominal surgery
  We will assess intraoperative transpulmonary pressure to evaluate respiratory mechanics during surgery.
Intraoperative respiratory system compliance | During abdominal surgery
  We will assess intraoperative respiratory system compliance to evaluate respiratory mechanics during surgery.
Intraoperative positive end-expiratory pressure (PEEP) levels | During abdominal surgery
  We will assess intraoperative PEEP values and their variability between patients and during surgery.

SECONDARY OUTCOMES:
Intraoperative gas exchange | During abdominal surgery
  We will assess intraoperative oxygenation and carbon dioxide elimination.
Plasma levels of biomarkers of lung injury | During abdominal surgery
  We will assess plasma concentrations of biomarkers of lung injury before and after surgery, including biomarkers of inflammation (interleukin-6, IL-6, interleukin-8, IL-8), epithelial injury (soluble form of the receptor for advanced glycation end-products, sRAGE, Club Cell protein-16, CC16), endothelial injury (angiopoietin-2, Ang-2), and endothelial-derived coagulation activation (plasminogen activator inhibitor-1, PAI-1).
Postoperative Pulmonary Complications | Within the first 7 postoperative days.
  We will assess the incidence and absolute number of postoperative pulmonary complications within the first 7 postoperative days.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Fernandez-Bustamante A, Sprung J, Parker RA, Bartels K, Weingarten TN, Kosour C, Thompson BT, Vidal Melo MF. Individualized PEEP to optimise respiratory mechanics during abdominal surgery: a pilot randomised controlled trial. Br J Anaesth. 2020 Sep;125(3):383-392. doi: 10.1016/j.bja.2020.06.030. Epub 2020 Jul 16. PMID 32682559